CLINICAL TRIAL: NCT01725087
Title: Efficacy, Safety, and Tolerability of GRT6005 in Subjects With Moderate to Severe Chronic Low Back Pain.
Brief Title: Efficacy and Safety of GRT6005 in Patients With Chronic Low Back Pain.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KF6005/06; 2012-001920-36 (EudraCT Number)
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Matching Placebo (Placebo Comparator): Twice daily oral administration of matching placebo for 14 weeks
  Interventions: Drug: Matching Placebo
- Low Dose GRT6005 (Experimental): Once daily GRT6005 low dose oral administration for 12 weeks with a titration period of 2 weeks.
  Interventions: Drug: Low Dose GRT6005
- Medium Dose GRT6005 (Experimental): Once daily GRT6005 medium dose oral administration for 12 weeks with a titration period of 2 weeks.
  Interventions: Drug: Medium Dose GRT6005
- High Dose GRT6005 (Experimental): Once daily GRT6005 high dose oral administration for 12 weeks with a titration period of 2 weeks.
  Interventions: Drug: High Dose GRT6005
- Tapentadol (Active Comparator): Twice daily oral administration of Tapentadol for 12 weeks with a titration period of 2 weeks.
  Interventions: Drug: Tapentadol

INTERVENTIONS:
Drug: Matching Placebo
  Arms: Matching Placebo
Drug: Low Dose GRT6005
  Arms: Low Dose GRT6005
Drug: Medium Dose GRT6005
  Arms: Medium Dose GRT6005
Drug: High Dose GRT6005
  Arms: High Dose GRT6005
Drug: Tapentadol
  Arms: Tapentadol

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of once daily orally administered GRT6005 in a total of 3 fixed doses compared to placebo in subjects with moderate to severe chronic Low Back Pain (LBP). The study includes a maximum of 21 days screening period followed by a 2-week titration period and 12-week maintenance double-blind treatment period and a 10-14 day safety follow up period. Patients who are eligible for the double-blind treatment period will be randomized to one of the following treatment groups: GRT6005 low-dose, GRT6005 medium dose, GRT6005 high-dose, Tapentadol or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low Back Pain of non-malignant origin and present for at least 3 months.
* Signed informed consent.
* Pain intensity score of 5 or greater on the 11-point numeric rating scale (where 0 indicates "no pain" and 10 indicates "as bad as you can imagine").
* On stable analgesic medications (non-opioid and/or opioid medications) for chronic low back pain with regular intake for at least 3 months and dissatisfied with current analgesic treatment.

Exclusion Criteria:

* Female subjects who are pregnant or are breastfeeding.
* Presence of risk factors for Torsade de Pointes.
* Any clinically significant disease or laboratory findings that may affect efficacy or safety assessments or may compromise the safety during trial participation, e.g., significant unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, metabolic, neurological, or psychiatric disorders.
* History of acute hepatitis within the past 3 months or chronic hepatitis or a positive result on anti-hepatitis A antibody, hepatitis B surface antigen, or anti-hepatitis C antibody. History of human immunodeficiency virus (HIV) infection.
* History of seizure disorder.
* Chronic low back pain potentially associated with a specific spinal cause.
* Surgery or painful procedure during or within 3 months of enrollment.
* Conditions that contribute and confound the assessment of pain.
* Subjects with impaired renal function.
* Subjects with impaired hepatic functionality.
* Neuromodulation.
* Cancer.
* Clinically relevant history of hypersensitivity, allergy or contraindications to any of the Investigational Medicinal Products' excipients, paracetamol/acetaminophen, tapentadol Hydrochloride, or opioid analgesics (or excipients).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1089 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
European Union: the change from baseline pain to the weekly average 24-hour pain during the entire 12 weeks of the maintenance phase of the double-blind Treatment Period. | Baseline to End of Treatment (Week 14)
United States: the change from baseline pain to the average 24-hour pain during Week 12 of the maintenance phase. | Baseline to End of Treatment (Week 14)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Chair — Grünenthal GmbH
Locations (79):
- Austria (5):
  - AT003, Senftenberg
  - AT004, Vienna
  - AT001, Vienna
  - AT005, Vienna
  - AT006, Vienna
- Belgium (3):
  - BE001, Brussels
  - BE002, Edegem
  - BE004, Genk
- Denmark (4):
  - DK004, Aalborg
  - DK001, Frederiksberg
  - Site DK002, Glostrup Municipality
  - DK003, Odense
- Finland (3):
  - FI005, Kokkola
  - FI001, Kuopio
  - FI003, Lahti
- Germany (16):
  - DE005, Bad Nauheim
  - DE014, Berlin
  - DE018, Berlin
  - DE011, Bochum
  - DE015, Böhlen
  - DE007, Dresden
  - DE016, Essen
  - DE001, Hamburg
  - DE006, Hamburg
  - DE008, Hanover
  - DE002, Leipzig
  - DE019, Leipzig
  - DE009, Mosbach
  - DE004, Munich
  - DE013, Rodgau
  - DE017, Wiesbaden
- Hungary (12):
  - HU010, Baja
  - HU008, Békéscsaba
  - HU011, Budapest
  - HU015, Budapest
  - HU005, Budapest
  - HU012, Budapest
  - HU003, Kecskemét
  - HU002, Kiskunfélegyháza
  - HU001, Makó
  - HU009, Nagykanizsa
  - HU014, Nyíregyháza
  - HU004, Szekszárd
- Netherlands (3):
  - NL003, Almere Stad
  - NL002, Eindhoven
  - NL005, Tiel
- Poland (16):
  - PL002, Elblag
  - PL015, Gdynia
  - PL006, Gdynia
  - PL001, Katowice
  - PL014, Katowice
  - PL008, Krakow
  - PL013, Krakow
  - PL011, Krakow
  - PL009, Lublin
  - PL016, Poznan
  - PL018, Poznan
  - PL012, Warsaw
  - PL004, Warsaw
  - PL010, Wroclaw
  - PL017, Wroclaw
  - PL005, Zgierz
- Spain (10):
  - ES004, A Coruña
  - ES002, Barcelona
  - ES006, Barcelona
  - ES001, Madrid
  - ES013, Madrid
  - ES008, Málaga
  - ES003, Oviedo
  - ES011, Oviedo
  - ES005, Santiago de Compostela
  - ES007, Seville
- Sweden (3):
  - SE001, Skene
  - SE002, Stockholm
  - SE004, Vällingby
- United Kingdom (4):
  - GB002, Liverpool
  - GB005, London
  - GB003, Manchester
  - GB004, Plymouth